CLINICAL TRIAL: NCT07143786
Title: Human Induced Neural Stem Cell-derived Exosomes for Treating Acute Ischemic Stroke: an Exploratory Clinical Trial
Brief Title: Human Induced Neural Stem Cell-derived Exosomes for Treating Acute Ischemic Stroke
Acronym: NSAIS
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Xuanwu Hospital, Beijing (Other)
Collaborators: Wiseheart Co.Ltd (Unknown)
Responsible Party: Principal Investigator, Junwei Hao, MD, Professor, Xuanwu Hospital, Beijing
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: iNSC-Exo-AIS2025
Record Dates: First submitted 2025-08-07; First posted 2025-08-27 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Ischemic Stroke, Acute
Keywords: induced neural stem cell; exosome; acute ischemic stroke; safety; efficacy
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exosome group (Experimental): Acute ischemic stroke patients that receive intravenous iNSC-Exo (5.0×10^11 ~ 2.0×10^12 particles) administration
  Interventions: Drug: iNSC-EV01
- Control group (Placebo Comparator): Acute ischemic stroke patients that receive intravenous placebo administration
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: iNSC-EV01 — Intravenous induced neural stem cell-derived exosome
  Arms: Exosome group
Drug: Placebo — iNSC-EV01 mimics
  Arms: Control group

SUMMARY:
A phase I/IIa clinical trial investigating the safety and preliminary efficacy of intravenous administration of human induced neural stem cell-derived exosomes for acute ischemic stroke

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-80 years (inclusive), regardless of gender;
2. Clinically diagnosed with an anterior circulation ischemic stroke in the current episode, confirmed by head MRI/CT, and able to receive the investigational product within 1 week after symptom onset;
3. National Institutes of Health Stroke Scale (NIHSS) score of 6-20 (inclusive) at randomization, with NIHSS item Ia score <2, and a change in NIHSS score from baseline to randomization of <4 points;
4. Female subjects of childbearing potential, or male subjects with partners of childbearing potential, must have no plans for pregnancy during the study and voluntarily use effective contraception;
5. Modified Rankin Scale (mRS) score of 0 or 1 before the onset of the current stroke symptoms, as self-reported or reported by family members.
6. All subjects, or their legal guardians, must provide written informed consent after receiving full information about the study and voluntarily participate in this clinical trial.

Exclusion Criteria:

1. Those with epilepsy, Alzheimer's disease, Parkinson's disease, severe depression, or other neurological disorders or psychiatric illnesses that the investigator deems would impair their ability to participate in the trial or affect the assessment of the study;
2. Patients who have experienced hemorrhagic transformation after the current ischemic stroke and are deemed unsuitable for participation in the clinical trial by the investigator;
3. Patients with malignant tumors, except for those with low-grade malignant tumors such as basal cell carcinoma, papillary thyroid carcinoma, and localized prostate cancer in situ, who have received radical treatment for more than five years;
4. Patients with severe infections, including sepsis, septic shock, severe pneumonia (refer to the 2007 criteria for severe pneumonia in adults by the Infectious Diseases Society of America/American Thoracic Society for the diagnosis of severe pneumonia);
5. Patients with respiratory failure, or those with current evidence of pulmonary embolism or suspected pulmonary embolism;
6. Patients whose organ function meets any one or more of the following criteria:

   1. Absolute Neutrophil Count (ANC) < 1.5 × 10⁹/L, Platelets (PLT) < 100 × 10⁹/L;
   2. Hemoglobin (Hb) < 90 g/L;
   3. Aspartate Aminotransferase (AST) > 2.5 × Upper Limit of Normal (ULN) and/or Alanine Aminotransferase (ALT) > 2.5 × ULN, Total Serum Bilirubin (TBIL) > 1.5 × ULN;
   4. Creatinine > 1.5 × ULN;
   5. For patients not receiving anticoagulant or antithrombotic therapy: International Normalized Ratio (INR) > 1.7 or Activated Partial Thromboplastin Time (APTT) > 1.25 × ULN; for patients receiving anticoagulant or antithrombotic therapy: INR > 3.0 or APTT > 1.5 × ULN;
7. Patients with a history of or current severe cardiovascular diseases:

   1. Those with myocardial ischemia, myocardial infarction, or unstable angina pectoris graded above CTCAE (Common Terminology Criteria for Adverse Events) Grade II;
   2. Severe arrhythmias deemed clinically significant by the investigator;
   3. Cardiac insufficiency of NYHA (New York Heart Association) Class III-IV;
   4. Those with other acute severe life-threatening complications;
8. Patients with poorly controlled hypertension (defined as persistent systolic blood pressure > 220 mmHg or diastolic blood pressure > 120 mmHg despite antihypertensive treatment);
9. Patients with poorly controlled diabetes mellitus (defined as blood glucose remaining > 16.8 mmol/L despite treatment) or hypoglycemia (blood glucose < 2.8 mmol/L);
10. Patients with a history of immunodeficiency, including: HIV-positive status, other acquired or congenital immunodeficiency diseases, idiopathic IgA deficiency, or those who have received systemic corticosteroid therapy (≥ 10 mg/day prednisone equivalent) or immunosuppressive drug therapy within 14 days prior to receiving the study drug, or who are expected to require such therapy during the trial;
11. Patients positive for Hepatitis B surface antigen (HBsAg) or Hepatitis B core antibody (HBcAb) with positive HBV-DNA, positive Hepatitis C antibody (HCV), or positive Treponema pallidum antibody (TPAb/RPR);
12. Patients who have participated in other drug clinical trials within 3 months prior to screening;
13. Patients with known allergies to the study drug or any of its components (e.g., human serum albumin);
14. Patients unable to undergo cranial CT/MRI examinations for any reason;
15. Patients who have undergone major surgery, suffered severe trauma within 3 months prior to the first dose, or plan to undergo surgery that may affect neurological function assessment during the trial;
16. Pregnant or lactating patients;
17. Patients with other severe systemic diseases, or a history of any diseases or laboratory abnormalities that may confound study results, interfere with the subject's participation in study procedures, or are not in the subject's best interest to participate, and who are deemed unsuitable for enrollment by the investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 38 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicity | Within 90 days
mRS | 90（±7）days
  modified Ranking Scale (mRS), ranging from 0 to 6, with higher scores indicating worse outcome, and a score of 6 representing death.

SECONDARY OUTCOMES:
AEs and SAEs | Within 90 days
  Adverse events and severe adverse events
mRS | 14（±1）days
  modified Ranking Scale (mRS), which ranges from 0 to 6, with higher scores indicating worse outcome, and a score of 6 representing death.
Percentage of mRS 0-2 | 14 (±1), 90 (±7) days
  modified Ranking Scale (mRS), which ranges from 0 to 6, with higher scores indicating worse outcome, and a score of 6 representing death.
NIHSS score change compared to baseline | 14 (±1), 90 (±7) days
  National Institutes of Health Stroke Scale (NIHSS), ranging from 0 to42, with higher score indicating more severe disabilities
Barthel Index change compared to baseline | 14 (±1), 90 (±7) days
  Barthel Index ranges from 0 to 100, with higher score indicating better daily living abilities
EQ5D-5L change compared to baseline | 14 (±1), 90 (±7) days
  EuroQol Five Dimensions Questionnaire (EQ5D) - Five levels, ranging from 5 to 25, with higher score indicating better outcome
Infarct volume change compared to baseline | 14 (±1), 90 (±7) days
  Infarct volume (cm3) measured by MRI

IPD SHARING:
Plan to Share IPD: No